CLINICAL TRIAL: NCT05611515
Title: Treatment of Supraglottic Squamous Cell Carcinoma With Advance Technologies: Observational Evaluation of Quality of Life, Oncological Outcomes, Functional Outcomes and Economical Resources
Brief Title: Treatment of Early Supraglottic Squamous Cell Carcinoma With Advance Technologies
Acronym: SUPRA-QoL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Principal Investigator, Professor Maximilien Gourdin, Professor, Centre Hospitalier Universitaire UCLouvain Namur
Other Study IDs: B0392022000044
Record Dates: First submitted 2022-10-14; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Supraglottic Squamous Cell Carcinoma; Early Stage (T1-T2, N0-N1,M0)
Keywords: Transoral Robotic Surgery (TORS); Transoral Laser Microsurgery (TLM); Intensity Modulated Radiation Therapy (IMRT); Early Squamous Cell Carcinoma; Supraglottic
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TORS: Patients operated by Trans-oral Robotic Surgery (TORS)
  Interventions: Procedure: TORS
- TLM: Patients operated by Trans-oral Laser Microsurgery (TLM)
  Interventions: Procedure: TORS
- IMRT: Patients treated by Intensity Modulated Radiation Therapy (IMRT)
  Interventions: Procedure: TORS

INTERVENTIONS:
Procedure: TORS — * Arm 1: Intensity-Modulated Radiation Therapy (IMRT)
  * Arm 2: Trans-oral Laser Microsurgery (TLM)
  * Arm 3: Trans-oral Robotic Surgery (TORS)
  Other Names: TLM; IMRT

SUMMARY:
In this project, the investigators will realize an observational, prospective, multicentric and international clinical trial, to objectively compare patients with SSCC according to 3 arms of treatment:

* Arm 1: Radiotherapy ± chemotherapy
* Arm 2: Trans-oral Laser Microsurgery (TLM)
* Arm 3: Trans-oral Robotic Surgery (TORS)

The main goal is to evaluate the efficacy of each treatment with four classes of outcomes:

* The quality of life (QoL) before and after each treatment option, using validated questionnaires
* Oncological outcomes
* Functional outcomes
* Economical Resources

The population will include cT1-T2 /cN0-N1/M0 supraglottic squamous cell carcinoma.

The primary outcome is a Clinical Dysphagia QoL evaluation assessed by the MD Anderson Dysphagia questionnaire. Secondary outcomes include others QoL evaluation, oncological and functional measures and cost parameters. The sample size needs to reach 36 patients per arm (total 108).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SSCC (with histological confirmation)

  * cT1-T2 / cN0-N1/ M0 according to 8th TNM classification (UICC/AJCC)
  * WITH a Multidisciplinary Tumor Board decision according to the NCCN or European guidelines
* Diagnostic imaging (Head and neck and pulmonary CT or PET/CT, +/- IRM if needed) realized within 1 month before the study inclusion
* ≥ 18 years old and able to provide an informed consent
* ECOG/WHO performance status ≤ 2

Exclusion Criteria:

* - Previous radiotherapy +/- chemotherapy treatment of the head and neck region
* Previous history of head and neck cancer within 5 years
* Prior invasive malignant disease unless disease-free for at least 5 years or more, with exception of non-melanoma skin cancer
* Non-supraglottic or unknown primary site
* Clinical and radiological signs of nodal extracapsular extension
* Significant trismus (maximum inter-incisal opening ≤ 35 mm)
* Pre-existing dysphagia not related to the cancer or the biopsy (from neurological disorders for example)
* Unable or unwilling to complete Quality of Life questionnaires
* Serious medical comorbidities or contraindication for surgery and/or radiation
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include cT1-T2 /cN0-N1/M0 supraglottic squamous cell carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Dysphagia QoL evaluation using MD Anderson Dysphagia Index (MDADI) | 1 year
  Clinical Dysphagia QoL evaluation after treatment will be assessed using MD Anderson Dysphagia Index (MDADI). MDADI consists of 20 items pooled in 4 subscales: the global scale (1 item); the functional scale (5 items); the physical scale (8 items); and the emotional scale (6 items). All items are scored on a 5-point scale (1-5), where "1" corresponds to "total agreement" and "5" to "total disagreement." All except 2 items were scored such that higher scores indicated higher functioning. Responses on all domains were summed to calculate the total score (MDADI-T). The maximum score is 100, indicating high functioning, and the minimum score is 20, indicating poor functioning.

SECONDARY OUTCOMES:
Quality of Life Measures with the validated European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire | baseline (before treatment), 3 - 6 - 9 - 12 - 18 - 24 months
  QoL will be evaluated with the validated European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire It is composed on five functional scales (physical, performance, cognitive, emotional and social), three symptoms scale (fatigue, pain, nausea and vomiting), a global health status/QoL scale and 6 simple items for assessment of symptoms or additional problems (dyspnea, loss of appetite, insomnia, financial difficulties, constipation and diarrhea). All of the scale and single item measures range in score from 0 to 100. Regarding functional and overall health status scales, higher scores relate to better quality of life; however, for the scales of symptoms, higher scores correspond to the higher presence of this symptom and, consequently, the worse quality of life.
Quality of Life Measures with the validated European Organization for Research and Treatment of Cancer (EORTC) H&N43 questionnaire | baseline (before treatment), 3 - 6 - 9 - 12 - 18 - 24 months
  QoL will be evaluated with the validated European Organization for Research and Treatment of Cancer (EORTC) H&N43 questionnaire It comprises 43 questions about symptoms and side effects of treatment, social function, body image and sexuality. It incorporates 12 symptom scales (pain, swallowing, problems with teeth, dry month and sticky saliva, problems with senses, speech, body image, social eating, sexuality, problems with shoulder, skin problems and fear of progression) and 7 simple items (problems opening mouth, coughing, social contact, swelling in the neck, weight loss, problem with wound healing and neurological problems). All of the scales and the single item measures range in score from 0 to 100. A high score represents a high level of symptomatology or problems.
Oncological Outcomes | 1 and 2 years
  Overall survival (%)
Oncological outcomes | 1 and 2 years
  Disease specific survival (%)
Oncological Outcomes | 1 and 2 years
  Disease-free survival (%)
Oncological Outcomes | 1 and 2 years
  Loco-regional recurrence rate (%)
Oncological Outcomes | 1 and 2 years
  Distant recurrence rate (%)
Functional Outcomes | baseline (before treatment), 1 - 3 - 6 - 9 - 12 - 18 - 24 months after treatment
  Swallowing function by FEES evaluation (Fiberoptic Endoscopic Evaluation of Swallowing) objectively evaluated by the Penetration-aspiration Scale (PAS) The PAS is an 8-point scale that rates the degree of airway invasion. Score of 1 is normal, score between 2-5 represent laryngeal penetration and scores up to 6 indicate airway aspiration.
Functional Outcomes | baseline (before treatment), 1 - 3 - 6 - 9 - 12 - 18 - 24 months after treatment
  Weight (Kilogrammes)
Functional Outcomes | baseline (before treatment), 1 - 3 - 6 - 9 - 12 - 18 - 24 months after treatment
  CTC-AE Score for early and late complication The Common Terminology Criteria for Adverse Events (CTC-AE) is a descriptive terminology which was published by the National Cancer Institute (NCI) as part of an ongoing effort to standardize adverse events (AE) reporting within oncology. AE are graded according to an ordinal scale where 1 represents asymptomatic or mild symptoms and 5 represents death from the AE. In between, 2 is moderate, 3 is severe, and 4 is life-threatening. E.g., with regard to dysphagia, the CTCAE uses the descriptive terminology listed in Table 1, columns 1 and 2. CTCAE dysphagia grades are based on symptoms, diet, and tube dependency. This scale will be filled in by the physician.
Functional Outcomes | 1 and 2 years
  Naso-gastric Feeding tube and/or gastrostomy use (duration in days)
Functional Outcomes | 1 and 2 years
  Tracheostomy use (duration in days)
Functional Outcomes | 1 and 2 years
  Need of hospitalization (yes or no; if yes, duration in days)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU UCL Namur, Yvoir, Namur, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hassid S, Krug B, Deheneffe S, Daisne JF, Delahaut G, Lawson G, Crott R, Van der Vorst S. Treatment of supraglottic squamous cell carcinoma with advanced technologies: observational prospective evaluation of oncological outcomes, functional outcomes, quality of life and cost-effectiveness (SUPRA-QoL). BMC Cancer. 2023 Jun 1;23(1):493. doi: 10.1186/s12885-023-10953-9. PMID 37264321